CLINICAL TRIAL: NCT02804932
Title: Nitrate Supplementation and Exercise Tolerance in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darren P Casey (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Darren P Casey, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201511802
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beetroot crystals (nitrate) (Experimental): Participants will receive a nitrate rich beetroot powder (10g/day) for 8 weeks.
  Interventions: Dietary Supplement: Super Beets
- Placebo (beetroot powder, no nitrate) (Placebo Comparator): Participants will receive a beetroot powder placebo (no nitrate) for 8 weeks.
  Interventions: Other: Super Beets Placebo

INTERVENTIONS:
Dietary Supplement: Super Beets — Nitrate rich beetroot powder (10g/day) for 8 weeks
  Other Names: Beetroot crystals
  Arms: Beetroot crystals (nitrate)
Other: Super Beets Placebo — Nitrate deficient beetroot powder (10g/day) for 8 weeks
  Other Names: Beetroot crystals no nitrate
  Arms: Placebo (beetroot powder, no nitrate)

SUMMARY:
The purpose of this study is to use a randomized, double-blind, placebo controlled study design to comprehensively investigate the impact of 8-weeks of dietary nitrate supplementation on skeletal muscle blood flow, mitochondrial function, and exercise capacity in patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Patients with type 2 diabetes (T2D) demonstrate a reduced exercise capacity, a powerful predictor of cardiovascular mortality, which may be due to reductions in skeletal muscle perfusion and mitochondrial dysfunction. Nitric oxide (NO) is a key molecule involved in in the regulation of blood flow to contracting muscles, as well as a critical mediator in mitochondrial respiration. However, there appears to be a decreased enzymatic synthesis of NO and an overall reduction of bioavailable NO in patients with T2D, which likely contributes to the reduced exercise capacity and tolerance. Accumulating evidence suggests that exogenous nitrate supplementation is an effective option for increasing NO bioavailability in vivo. The purpose of the proposal is to use a randomized, double-blind, placebo controlled study design to comprehensively investigate the impact of 8-weeks of dietary nitrate supplementation on skeletal muscle blood flow, mitochondrial function, and exercise capacity in patients with T2D. The central hypothesis is that increasing NO bioavailability via dietary nitrate supplementation in patients with T2D will lead to improved oxygen delivery and utilization during exercise. To address this hypothesis a highly mechanistic and translational experimental strategy will be used to explore whether increased NO bioavailability via dietary nitrate supplementation improves skeletal muscle perfusion during exercise (Aim 1), enhances mitochondrial biogenesis and function (Aim 2), and improves exercise capacity and efficiency (Aim 3). Collectively, these studies will provide important mechanistic insight into the therapeutic potential of dietary nitrate supplementation for improving skeletal muscle blood flow, mitochondrial function and exercise capacity in patients with T2D.

ELIGIBILITY:
For 50 patients with documented Type 2 diabetes

Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is > or = 40 and < or = 77 years of age
* Documented Type 2 diabetes

Exclusion Criteria:

* diagnosis of type 2 diabetes < 3 years prior to enrollment
* HbA1c <6.0% or >10.0%
* body mass index > 42 kg/m2
* incident cardiovascular events in the last year (heart attack, stroke)
* symptomatic coronary artery disease and/or heart failure
* uncontrolled hypertension
* hypotension (resting systolic BP < 90 mmHg)
* renal impairment with creatinine clearance (eGFR) of <50 ml/min
* smoking or history of smoking within past one year
* use of medication which contain nitrates
* use of anti-coagulant drugs
* use of anti-platelet drugs
* participation in research studies in which medications or interventions are given which would potentially alter subject responses in the current study

For 15 age- and weight-matched nondiabetic control subjects

Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is > or = 40 and < or = 77 years of age

Exclusion Criteria:

* Diagnosis of diabetes (Type 1 or Type 2)
* body mass index > 42 kg/m2
* incident cardiovascular events in the last year (heart attack, stroke)
* symptomatic coronary artery disease and/or heart failure
* uncontrolled hypertension
* hypotension (resting systolic BP < 90 mmHg)
* renal impairment with creatinine clearance (eGFR) of <50 ml/min
* smoking or history of smoking within past one year
* use of medication which contain nitrates
* use of anti-coagulant drugs
* use of anti-platelet drugs
* participation in research studies in which medications or interventions are given which would potentially alter subject responses in the current study

Ages: 40 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren P Casey, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bock JM, Hanson BE, Miller KA, Seaberg NT, Ueda K, Feider AJ, Hanada S, Lira VA, Casey DP. Eight weeks of inorganic nitrate/nitrite supplementation improves aerobic exercise capacity and the gas exchange threshold in patients with type 2 diabetes. J Appl Physiol (1985). 2022 Dec 1;133(6):1407-1414. doi: 10.1152/japplphysiol.00478.2022. Epub 2022 Nov 3. PMID 36326473
- [Derived] Bock JM, Hughes WE, Ueda K, Feider AJ, Hanada S, Casey DP. Dietary Inorganic Nitrate/Nitrite Supplementation Reduces Central and Peripheral Blood Pressure in Patients With Type 2 Diabetes Mellitus. Am J Hypertens. 2022 Sep 1;35(9):803-809. doi: 10.1093/ajh/hpac068. PMID 35639721

RESULTS

PARTICIPANT FLOW:
Groups:
- Nondiabetic Control Subjects: All pre supplementation measures and study visits will be performed in a group of 15 nondiabetic control subjects to allow us to 1) quantify the degree of impairment in T2D prior to intervention and 2) assess the effectiveness of the nitrate therapy in restoring the primary outcome measures back to 'normal'. Nondiabetic controls will not receive an 8-week beetroot supplementation.
Period: Overall Study
Arm/Group | Beetroot Crystals (Nitrate) | Placebo (Beetroot Powder, no Nitrate) | Nondiabetic Control Subjects
Started | 20 | 19 | 15
Completed | 19 | 18 | 15
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beetroot Crystals (Nitrate) | Placebo (Beetroot Powder, no Nitrate) | Nondiabetic Control Subjects | Total
Number analyzed (Participants) | 20 | 19 | 15 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 11 | 37
  >=65 years | 8 | 5 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.7) | 58.7 (8.8) | 60.2 (9.2) | 59.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 15 | 14 | 10 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Maximal Exercise Capacity (VO2max)
Description: A 12-lead ECG, symptom limited cardiopulmonary exercise testing with gas exchange measurements will be performed on a cycle ergometer using a ramp protocol to determine maximal aerobic capacity (VO2max) and exercise efficiency.
Time Frame: Pre and post 8 weeks of dietary nitrate supplementation
Population: One subject in the nitrate group did not reach maximal criteria during testing. Therefore, VO2max data was analyzed only in 18 participants in the nitrate group. Nondiabetic control subjects only completed VO2max testing once (same time point as pre measurements for T2D subjects).
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Beetroot Crystals (Nitrate) | Placebo (Beetroot Powder, no Nitrate) | Nondiabetic Control Subjects
Number analyzed (Participants) | 18 | 18 | 15
mL/kg/min
  VO2max - Pre supplementation | 20.7 (7.0) | 20.0 (4.2) | 27.6 (8.7)
  VO2max - Post supplementation: number analyzed (Participants) | 18 | 18 | 0
  VO2max - Post supplementation | 21.9 (7.4) | 19.7 (4.6) |

2. Primary Outcome: Change in Skeletal Muscle Perfusion During Exercise
Description: Forearm blood flow will be determined using Doppler ultrasound during rhythmic forearm exercise.
Time Frame: Pre and post 8 weeks of dietary nitrate supplementation
Population: Nondiabetic control subjects only completed rhythmic forearm exercise and forearm blood flow measurements at one study visit (same time point as pre measurements for T2D subjects).
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Beetroot Crystals (Nitrate) | Placebo (Beetroot Powder, no Nitrate) | Nondiabetic Control Subjects
Number analyzed (Participants) | 19 | 18 | 15
ml/min
  Forearm Blood Flow - pre supplementation | 156 (69) | 143 (69) | 200 (64)
  Forearm Blood Flow - post supplementation: number analyzed (Participants) | 19 | 18 | 0
  Forearm Blood Flow - post supplementation | 175 (73) | 143 (66) |

3. Primary Outcome: Change in Skeletal Muscle Mitochondrial Function
Description: Muscle biopsies were obtained from the vastus lateralis using a Bergstrom needle with suction under local anesthesia, which will yield ~200-250mg of tissue. Mitochondrial function was assessed as follows: Fiber bundles were chemically permeabilized with saponin and mitochondrial respiration was analyzed by in situ high-resolution respirometry at 37°.
Time Frame: Pre and post 8 weeks of dietary nitrate supplementation
Population: Final number of participants studied with muscle biopsies was smaller than the total number of subjects enrolled in the study. The lower number was influenced by: (i) subjects not consenting to the muscle biopsy procedure; or (ii) technical problems (ex: not enough muscle tissue and/or extensive proportion of intramuscular fat obtained).
  Nondiabetic control subjects only had muscle biopsies performed at one time point (same time point as pre measurements for T2D subjects).
Measure: Mean (Standard Deviation); unit: Oxygen Flux, JO2 (pmol/(s*mg))
Arm/Group | Beetroot Crystals (Nitrate) | Placebo (Beetroot Powder, no Nitrate) | Nondiabetic Control Subjects
Number analyzed (Participants) | 12 | 6 | 10
Oxygen Flux, JO2 (pmol/(s*mg))
  CHO-supported respiration - Pre | 64.6 (22.2) | 71.0 (20.5) | 87.5 (21.5)
  CHO-supported respiration - Post: number analyzed (Participants) | 12 | 6 | 0
  CHO-supported respiration - Post | 75.4 (16.4) | 59.8 (11.1) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration each subject was enrolled in the study, which was up to 12 weeks.
Arm/Group | Beetroot Crystals (Nitrate) | Placebo (Beetroot Powder, no Nitrate) | Nondiabetic Control Subjects
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/15

LIMITATIONS AND CAVEATS:
Final number of participants studied with muscle biopsies was smaller than the total number of subjects enrolled in the study. The lower number was influenced by: (i) subjects not consenting to the muscle biopsy procedure; or (ii) technical problems occurring in at least one of the testing visits (ex: not enough muscle tissue and/or extensive proportion of intramuscular fat obtained).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT02804932/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT02804932/SAP_001.pdf